CLINICAL TRIAL: NCT00607204
Title: Neurobiology of Individual Differences in Sleep Duration
Brief Title: Examining the Biological Factors That Affect Sleep Duration
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Daniel Aeschbach, Associate Neuroscientist, Brigham and Women's Hospital
Other Study IDs: 559; R01HL077399 (NIH)
Record Dates: First submitted 2008-02-04; First posted 2008-02-05 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Sleep; Circadian Rhythm; Cognitive Performance
Keywords: Basic Research; Individual Sleep Duration; Melatonin; Electroencephalogram; Alertness; Mood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Sleep is necessary for healthy functioning, and people who sleep too little or too much may have an increased risk of developing health problems. This study will examine people who regularly sleep for short or long amounts of time to understand the biological factors that determine how much sleep a person needs.

DETAILED DESCRIPTION:
The amount of sleep people require depends on many factors, including age, but experts agree that most adults need 7 to 8 hours of sleep a night. People who sleep for shorter or longer amounts of time may be at risk of developing memory problems, heart disease, obesity, and diabetes. The duration and timing of sleep are regulated by an interaction between the circadian pacemaker, or biological clock, and the sleep homeostat, which is an internal account of the amount of sleep a person has received recently. It is unknown whether there is a biological or genetic basis for the amount of sleep a person needs. This inpatient study will examine two extreme sleep groups: short sleepers who sleep 6.5 or less hours a night and long sleepers who sleep 9 or more hours a night. Participants will be exposed to identical sleep opportunities and living conditions. Using hormone analysis to examine participants' circadian rhythms, researchers will evaluate the biological differences that people undergo during the sleep process. Results from this study may help researchers understand whether sleep duration and sleep needs differ among people because of biological and genetic variations.

Over a period of 4 to 6 weeks, potential study participants will attend 4 to 6 screening visits, which will include a medical history review, physical exam, blood and urine collection, electrocardiogram (EKG) to measure electrical activity of the heart, a psychological assessment, and an overnight stay in a sleep laboratory. For 3 weeks, potential participants will also wear an activity monitor, and they will record sleep habits electronically and in a daily diary.

Participants who are eligible for the study will spend 28 days in the Intensive Physiological Monitoring Unit of the Clinical and Translational Sciences Center at the Brigham and Women's Hospital. Participants will not have access to a clock, radio, television, or computer, and they will not be allowed any outside contact. Most days participants will remain in bed for 10 to 14 hours; however, at selected times during the study, participants will remain inactive for periods of 32 to 64 hours and will stay awake for 32 to 40 hours. Throughout the study, participants' sleep patterns will be monitored continuously by a wrist activity recorder. Heart rhythms, brain electrical activity, eye movements, and temperature will also be measured continuously. At different times throughout the study, participants will undergo urine, saliva, and blood collection; alertness, mood, and performance evaluations; and blood pressure measurements. Upon release from the research center, participants will maintain a sleep diary for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Routinely sleeps 6.5 hours or less a night, or routinely sleeps 9 hours or more a night
* In good health

Exclusion Criteria:

* Diagnosed with a sleep disorder
* Currently uses medications
* Performed night shift work in the 3 years before study entry
* History of psychiatric illness

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will include healthy people who are catagorized as either short sleepers or long sleepers.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2005-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm assessment based on plasma melatonin and other hormones; sleep and EEG analysis; measurements of cognitive performance, alertness, and mood | Measured during the 4-week inpatient stay

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Aeschbach, PhD, Principal Investigator — Brigham & Women's Hospital, Boston, MA
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Aeschbach D, Sher L, Postolache TT, Matthews JR, Jackson MA, Wehr TA. A longer biological night in long sleepers than in short sleepers. J Clin Endocrinol Metab. 2003 Jan;88(1):26-30. doi: 10.1210/jc.2002-020827. PMID 12519823
- [Background] Aeschbach D, Postolache TT, Sher L, Matthews JR, Jackson MA, Wehr TA. Evidence from the waking electroencephalogram that short sleepers live under higher homeostatic sleep pressure than long sleepers. Neuroscience. 2001;102(3):493-502. doi: 10.1016/s0306-4522(00)00518-2. PMID 11226688
- [Background] Aeschbach D, Cajochen C, Landolt H, Borbely AA. Homeostatic sleep regulation in habitual short sleepers and long sleepers. Am J Physiol. 1996 Jan;270(1 Pt 2):R41-53. doi: 10.1152/ajpregu.1996.270.1.R41. PMID 8769783
- See also: Click here for the Division of Sleep Medicine at Harvard Medical School Web site — http://sleep.med.harvard.edu/